CLINICAL TRIAL: NCT05865067
Title: Yoga Therapy for Latino Preschool Children With Oppositional Defiant Behaviors
Brief Title: Yoga Therapy and Oppositional Defiant Disorder Behaviors
Acronym: YTODD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Puerto Rico (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency); American Psychiatric Association (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2290034907
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-05

CONDITIONS: Oppositional Defiant Disorder in Children; Oppositional Defiant Disorder
Keywords: yoga; yoga therapy; preschool; odd; oppositional defiant disorder; latino; children
MeSH Terms: conditions — Oppositional Defiant Disorder | interventions — Yoga; Exercise

STUDY DESIGN:
Intervention Model Description: This is a Pilot efficacy, randomized intervention, wait-list controlled clinical trial to evaluate the feasibility of Yoga Therapy for Latino Preschool children aged 4 to 6 years old with ODD. This design makes it comparable to the pilot efficacy study done in the same age and diagnostic group by Dr. Matos, which evaluated PCIT efficacy. We will recruit participants by flyers to obtain 34 patients and 68 parents; after confirming ODD trait with DBRS, they will be randomized to intervention and wait-list control groups. Randomization will be performed in a 3:2 ratio (Yoga-Therapy: Wait-List; 21:13). Flyers, newspapers, radio, and television ads will recruit participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Therapy (Experimental): Participation will consist of 1) a telephone survey to screen for exclusion factors; 2) filling out two questionnaires and consent at the first visit; 3) filling out four questionnaires on orientation day (day 2); 4) receiving an orientation for you and your child and receive an educational pamphlet on the 2nd and 15th (closing); 5) participate in the 12 Yoga sessions with your child (Saturdays) with a weekly call to remind you of your appointment; 6) fill out a questionnaire on day 8 (6th yoga class); 7) fill out five questionnaires on the 15th (closing); 8) a possible assessment of your child's heartbeat at the 12 intervention sessions (will be randomly selected); 9) an evaluation of your child's sweating at the first visit (orientation) and at visit 15 (closing); 10) a last visit to finish and offer additional information (day 15; closing); 11) a telephone survey three months (day 16) after completing the study.
  Interventions: Other: Yoga Therapy
- Wait-List with Exercise (Active Comparator): Participation consists of 1) a telephone survey to screen for exclusion factors; 2) filling out two questionnaires and informed consent at the first visit; 3) filling out four questionnaires in the second meeting (day 2 of orientation); 4) filling out six questionnaires in the last meeting (day 15; closure); 4) receive a 30-45 minute video orientation and psychoeducation (where you will also receive an educational brochure) and a series of exercise recommendations for you and your child on day 2 (orientation); 5) 12 phone calls (once a week); 6) an evaluation of your child's sweating at the first visit (orientation) and last visit (day 15; closure); 7) an evaluation of your child's heart rhythm at the first visit (orientation) and last visit (day 15; closure); 8) a telephone survey (day 16; follow-up) 3 months after completing the study; 9) a call at the end of the study to coordinate the Yoga sessions for you and your child once the first group has finished.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Yoga Therapy — The intervention sessions will consist of 12 yoga therapy sessions, each one approximately 30 to 45 minutes long, it will be given once a week (on Saturdays) in a room in the building of the School of Health Professions in the Campus of Medical Sciences from the University of Puerto Rico.
  Arms: Yoga Therapy
Other: Exercise — The wait-list control group will be motivated to exercise at home (except for Yoga).
  Arms: Wait-List with Exercise

SUMMARY:
This clinical trial aims to learn about, test, and compare the effect yoga therapy has on improving disruptive behaviors (e.g., oppositional defiant disorder) in Latino preschool children and parent-child interactions.

The main question[s] it aims to answer are:

* Can Yoga Therapy improve disruptive behaviors in Latino preschool children with Oppositional Defiant Disorder traits?
* Can Yoga Therapy improve parent-child interactions in Latino preschool children with Oppositional Defiant Disorder traits?

Participants will:

* Complete an initial survey to screen for inclusion and exclusion factors
* Fill out two questionnaires and consent form at the first visit
* Fill out four questionnaires on orientation day (day 2)
* Receive orientation and receive an educational pamphlet on the 2nd and 15th (closing) days
* Participate in the 12 Yoga sessions with a weekly call to remind them of their appointment
* Fill out a questionnaire on day 8 (6th yoga class)
* Fill out five questionnaires on the 15th (closing)
* Receive a possible assessment of the child's heartbeat at the 12 intervention sessions (will be randomly selected) with a heart rate variability monitor
* Receive an evaluation of the child's sweating at the first visit (orientation) and visit 15 (closing)
* Participate in a last visit to finish and offer additional information (day 15; closing)
* Participate in a telephone survey three months (day 16) after completing the study.

Control group participation will consist of:

* Fill a telephone survey to screen for inclusion and exclusion factors
* Fill out two questionnaires and informed consent at the first visit
* Fill out four questionnaires in the second meeting (day 2 of orientation)
* Fill out six questionnaires in the last meeting (day 15; closure)
* Receive a 30-45 minute video orientation and psychoeducation (where they will also receive an educational brochure) and a series of exercise recommendations for parent and children on day 2 (orientation)
* Receive 12 phone calls (once a week) to remind them to exercise and evaluate if they exercised the week before
* Receive an evaluation of the child's sweating at the first visit (orientation) and last visit (day 15; closure)
* Receive an evaluation of the child's heart rhythm at the first visit (orientation) and last visit (day 15; closure)
* Fill out a telephone survey (day 16; follow-up) three months after completing the study
* Receive a call at the end of the study to coordinate the Yoga sessions for parents and children once the intervention group has completed their participation.

Researchers will compare Yoga therapy to exercise to see if there is a change in disruptive behaviors and parent-child interactions.

DETAILED DESCRIPTION:
In the process of obtaining the 34 participants and their respective fathers/mothers, they will be randomly divided between the two possible groups (YogaTherapy or Psycho-Education). This will be done through the recruitment process as follows: the first child listed will go to the intervention group, the second to the waiting list, the third to the intervention, the fourth to the waiting list, and so on. The same will be done for the girls: the first to the intervention group, the second to the waiting list, etc.

The intervention group:

In the first face-to-face meeting, you will complete five questionnaires [Your Child's Medical History, Disruptive Behavior Scale, Parenting Questionnaire-Preschool Edition, Parent Stress Index-Short Version, Sense of Parenting]. You will do a baseline assessment of your child's heartbeat and sweating. Once the intervention sessions begin, they will participate in 12 sessions, each approximately 30 to 45 minutes long, which will occur once a week (on Saturdays) in a room in the School of Health Professions building at the Medical Sciences Campus of the University of Puerto Rico. Later on, you will be told the room and the floor where you are staying and where you will receive the intervention: it will always be the same day, at the same time.

* In 12 sessions, the child's heart rate will be evaluated with a monitor that will be placed on his ear (this measurement will only be done to one child out of the possible five who will be taking his session. It will be determined randomly which child will receive an evaluation of your heart rhythm)
* In 4 sessions, you will complete the DBRS questionnaire (disruptive behavior scale - Spanish version).
* In the first session, you will fill out five questionnaires [Your Child's Medical History, Disruptive Behaviors Scale, Parenting Questionnaire-Preschool Edition, Parenting Stress Index-Short Version, Sense of Parenting] and assess your child's heart rate and sweating
* In the last session, you will complete five questionnaires [Disruptive Behavior Scale, Parenting Questionnaire-Preschool Edition, Parent Stress Index-Short Version, Sense of Competence as a Parent, Assessment of Therapy Offered] and assess your heart rate and your child's sweating one last time. Sweating will be measured with a machine where a Velcro ring will be placed on the ring finger of your non-right hand.
* You must wear a mask at all times. All staff will be wearing a mask at all times. Products will be disinfected with chlorine before and after each session.

Your total participation in the study (in the intervention group) will consist of 3 face-to-face months (one Saturday a week) up to a total of 6 months and 3 weeks if we include orientation day, closing day, and the call at 3 months after completing the study.

The control group:

* In the first face-to-face meeting, you will fill out six questionnaires [Your Child's Medical History, Disruptive Behaviors Scale, Parenting Questionnaire-Preschool Edition, Parenting Stress Index-Short Version, Sense of Competence as a Parent, Evaluation of therapy offered] and a baseline assessment of your child's heartbeat and sweating will be done.
* In 3 sessions, you will complete the DBRS questionnaire (disruptive behavior scale - Spanish version).
* In the first session, you will fill out five questionnaires [Your Child's Medical History, Disruptive Behaviors Scale, Parenting Questionnaire-Preschool Edition, Parenting Stress Index-Short Version, Sense of Parenting] and assess your child's heart rate and sweating
* In the last session, you will fill out five questionnaires [Disruptive Behavior Scale, Parenting Questionnaire-Preschool Edition, Parent Stress Index-Short Version, Sense of Competence as a Parent, Assessment of Therapy Offered], and we will assess your heart rate and your child's sweating one last time. Sweating will be measured with a machine where a Velcro ring will be placed on the ring finger of your non-right hand.

Their total participation in the study (in the waiting list group) consists of 3 face-to-face weeks - for the screening day, orientation day, and closing day up to a total of 6 months, considering the call 3 months after finishing the study.

This is an experimental study where the Yoga intervention will be compared with the waiting list (control group), and Yoga Therapy will be compared to Psychoeducation. To participate in our study, you have to give permission to videotape the sessions. Each session will be recorded with video to improve the intervention, to be able to transcribe the ideas expressed (anonymously), control the quality of each intervention and ensure the fidelity of the instructors to the manual; each recording will be labeled with your identifier code, without any personal information that can identify you or your child. Once the investigation is completed, the recordings will be kept for five years at the Center for the Study and Treatment of Fear and Anxiety (CETMA) under the custody of Dr. Karen Martínez in office 236 of the Health Professions Studies Building at the Medical Sciences Campus of the University of Puerto Rico. Electronic and paper data will be stored in the mentioned office for five years. Electronic data will be erased after five years, and the hard drive will be formatted after erasing the data. Data on paper is shredded.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 4 to 6 years
* The child has oppositional defiant disorder (ODD) traits
* The child is not under pharmacological treatment for oppositional defiant disorder (ODD)

Exclusion Criteria:

* The child has speech or hearing problems
* The child has a history of developmental disorders (severe)
* The child is using pharmacotherapy - psychoactive medications
* Parents are not willing to put psychological treatments on hold while they are in this study
* The child is or has received training in yoga
* The parents, legal guardians, or the person in charge have problematic use of substances.
* There is a history of mental or physical abuse in the home [If identified, the referral protocol will be activated]
* The child is less than four years old or older than six years old

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Disruptive Behavior Disorder Rating Scale (DBRS) | 15 weeks
  The Disruptive Behavior Scale for Children (DBRS; Spanish Version), is used as a screening and outcome measure. The DBRS will be administered to the intervention and control groups at Day 1, Day 8, Day 14, Day 15, and Day 16 (3-month follow-up). This scale has 41 DSM items on a 4-point scale, answer options include: never or rarely, sometimes, often, or very often, ranging from 0 to 3 points, respectively, using the past six months as a time frame. A total of 3 or more items (DBRS-ODD) must be marked as "often" or "very often" by parents to meet the inclusion criteria for an ODD trait. The outcome for DBRS is a change from baseline levels between two groups after adjusting for baseline measurements. Dr. Russel Barkley authorized the use of this instrument (Spanish Version).

SECONDARY OUTCOMES:
Alabama Parenting Questionnaire Preschool Version (APQ-Pr) | 15 weeks
  The APQ is a 42-item self-report measure of parenting characteristics, which have been associated with disruptive behaviors for children 6 to 13 years of age. The items are categorized into five subscales reflective of parenting practices; Parents report how frequently they use the described parenting strategies: positive parental involvement, positive parenting discipline techniques, poor monitoring/supervision, inconsistent discipline, and corporal punishment; items are rated on a 5-point Likert-scale (1 = Never to 5 = Always). Various studies have tested the scale reliability; internal consistency for all scales ranges from .80 to .46, while temporal stability ranges from .89 to .6929,30,39. Alpha scores range from .86 to .5429. There is a Spanish version available. Clerkin et al. (2007) adapted this instrument for Preschool children (APQ-Pr).
Parenting Stress Index, Short Form (PSI-SF) | 15 weeks
  Parenting Stress Index, Short Form (PSI-SF) measures parenting stress via a 36-item self-report measure. Parents report their agreement with each statement in a 5-point Likert Scale ("Strongly Agree" to "Strongly Disagree") regarding three subscales (Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child), a Defensive Responding Scale, and Total Score. Both tools will be administered on Day 2 (Orientation) and Day 15 (Closure) for both intervention and control groups. The outcome for APQ-Pr and PSI-SF is a change from baseline levels between the two groups after adjusting for baseline measurements. PSI-SF instrument is freely available online. The use of the APQ-Pr instrument (Spanish Version) was authorized by Nuria de la Osa.
Parent Sense of Competence Scale (PSOC) | 15 weeks
  Trained personnel will evaluate parental satisfaction, and efficacy will be measured with the Parent Sense of Competence Scale (PSOC) its two subscales are "Satisfaction", which evaluates parental frustration, anxiety, and motivation as an affective dimension while "Efficacy" evaluates competence, problem-solving ability, and parenting role capability as an instrumental dimension. PSOC is a 17-item report measure that responded to a 6-point Likert Scale (from 1 = Strongly Agree to 6 = Strongly Disagree). Nine items are reverse scaled (i.e., higher scores indicate a lower parental sense of competence). A higher score for Total Score indicates a higher parenting sense of competence. Test and retest reliability ranges from .46 to .82, and alpha levels range from .82 to .7034,35. PSOC tools will be administered on Day 2 (Orientation) and Day 15 (Closure) for both intervention and control groups.
Therapy Evaluation Scale (TES) | 15 weeks
  The therapy Evaluation Scale (TES) evaluates perceived parental satisfaction with treatment, the ability to adequately apply treatment strategies at home, quality of the therapist-client relationship, and asks if the client has any suggested changes to improve the treatment. Our collaborator developed this scale for Puerto Rican families in 1997 (Matos, 1997), and it was adapted to ensure relevance to Yoga Therapy. The design of the items does not allow an analysis of psychometric properties. The TES tool will be administered on Day 15 (Closure) for both intervention and control groups. The outcome for PSOC is a change from baseline levels between two groups after adjusting for baseline measurements. PSOC is freely available online. Dr. Maribel Matos authorized the use of this TES (Spanish Version).
Heart rate variability (HRV) | 15 weeks
  We will measure heart rate variability (HRV) pre- and post-intervention in both groups with the Inner Balance Bluetooth BT4.0 (BLE-Bluetooth Low energy) monitor, which works at an output power range of 0.5 milliwatts (mW) or less. HRV will be recorded as described by McCraty et al. (2009, p.23). Baseline HRV will be measured, at the beginning of each session. The monitor is placed on the child's earlobe and transmits via Bluetooth. The HeartMath quantifies heart rhythm by identifying the maximum peak in the 0.04-0.26 Hz range26. The methodology of the HeartMath is described by McCraty et al. (2009, p.23)26. HR will be measured during pre- and post-yoga therapy sessions in a randomly selected family unit; one child of a family unit per intervention day will receive HRV measurements. Dr. Esparham will be a consultant.

CONTACTS AND LOCATIONS:
Overall Officials: Karen G Martínez, MD, MSc, Principal Investigator — University of Puerto Rico Department of Psychiatry
Locations (1):
- University of Puerto Rico Medical Sciences Campus, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stormshak EA, Bierman KL, McMahon RJ, Lengua LJ. Parenting practices and child disruptive behavior problems in early elementary school. Conduct Problems Prevention Research Group. J Clin Child Psychol. 2000 Mar;29(1):17-29. doi: 10.1207/S15374424jccp2901_3. PMID 10693029
- [Background] Canino G, Shrout PE, Rubio-Stipec M, Bird HR, Bravo M, Ramirez R, Chavez L, Alegria M, Bauermeister JJ, Hohmann A, Ribera J, Garcia P, Martinez-Taboas A. The DSM-IV rates of child and adolescent disorders in Puerto Rico: prevalence, correlates, service use, and the effects of impairment. Arch Gen Psychiatry. 2004 Jan;61(1):85-93. doi: 10.1001/archpsyc.61.1.85. PMID 14706947
- [Background] Steiner H, Remsing L; Work Group on Quality Issues. Practice parameter for the assessment and treatment of children and adolescents with oppositional defiant disorder. J Am Acad Child Adolesc Psychiatry. 2007 Jan;46(1):126-141. doi: 10.1097/01.chi.0000246060.62706.af. PMID 17195736
- [Background] Matos M, Bauermeister JJ, Bernal G. Parent-child interaction therapy for Puerto Rican preschool children with ADHD and behavior problems: a pilot efficacy study. Fam Process. 2009 Jun;48(2):232-52. doi: 10.1111/j.1545-5300.2009.01279.x. PMID 19579907
- [Background] Tyagi A, Cohen M. Yoga and heart rate variability: A comprehensive review of the literature. Int J Yoga. 2016 Jul-Dec;9(2):97-113. doi: 10.4103/0973-6131.183712. PMID 27512317
- [Background] Herbert A, Esparham A. Mind-Body Therapy for Children with Attention-Deficit/Hyperactivity Disorder. Children (Basel). 2017 Apr 25;4(5):31. doi: 10.3390/children4050031. PMID 28441363
- [Background] Schoorl J, Van Rijn S, De Wied M, Van Goozen SH, Swaab H. Variability in emotional/behavioral problems in boys with oppositional defiant disorder or conduct disorder: the role of arousal. Eur Child Adolesc Psychiatry. 2016 Aug;25(8):821-30. doi: 10.1007/s00787-015-0790-5. Epub 2015 Nov 25. PMID 26608403
- [Background] Bauermeister JJ, Puente A, Martinez JV, Cumba E, Scandar RO, Bauermeister JA. Parent perceived impact of Spaniard boys' and girls' inattention, hyperactivity, and oppositional defiant behaviors on family life. J Atten Disord. 2010 Nov;14(3):247-55. doi: 10.1177/1087054709347180. Epub 2009 Sep 18. PMID 19767594
- [Background] Harvey EA, Youngwirth SD, Thakar DA, Errazuriz PA. Predicting attention-deficit/hyperactivity disorder and oppositional defiant disorder from preschool diagnostic assessments. J Consult Clin Psychol. 2009 Apr;77(2):349-54. doi: 10.1037/a0014638. PMID 19309194
- [Background] Lahey BB, Pelham WE, Stein MA, Loney J, Trapani C, Nugent K, Kipp H, Schmidt E, Lee S, Cale M, Gold E, Hartung CM, Willcutt E, Baumann B. Validity of DSM-IV attention-deficit/hyperactivity disorder for younger children. J Am Acad Child Adolesc Psychiatry. 1998 Jul;37(7):695-702. doi: 10.1097/00004583-199807000-00008. PMID 9666624
- [Background] Loeber R, Burke JD, Lahey BB, Winters A, Zera M. Oppositional defiant and conduct disorder: a review of the past 10 years, part I. J Am Acad Child Adolesc Psychiatry. 2000 Dec;39(12):1468-84. doi: 10.1097/00004583-200012000-00007. PMID 11128323
- [Background] Canino G, Polanczyk G, Bauermeister JJ, Rohde LA, Frick PJ. Does the prevalence of CD and ODD vary across cultures? Soc Psychiatry Psychiatr Epidemiol. 2010 Jul;45(7):695-704. doi: 10.1007/s00127-010-0242-y. Epub 2010 Jun 9. PMID 20532864
- [Background] Speltz ML, McClellan J, DeKlyen M, Jones K. Preschool boys with oppositional defiant disorder: clinical presentation and diagnostic change. J Am Acad Child Adolesc Psychiatry. 1999 Jul;38(7):838-45. doi: 10.1097/00004583-199907000-00013. PMID 10405501
- [Background] Burke JD, Waldman I, Lahey BB. Predictive validity of childhood oppositional defiant disorder and conduct disorder: implications for the DSM-V. J Abnorm Psychol. 2010 Nov;119(4):739-51. doi: 10.1037/a0019708. PMID 20853919
- [Background] Jensen PS, Kenny DT. The effects of yoga on the attention and behavior of boys with Attention-Deficit/ hyperactivity Disorder (ADHD). J Atten Disord. 2004 May;7(4):205-16. doi: 10.1177/108705470400700403. PMID 15487477
- [Background] Hagen I, Nayar US. Yoga for Children and Young People's Mental Health and Well-Being: Research Review and Reflections on the Mental Health Potentials of Yoga. Front Psychiatry. 2014 Apr 2;5:35. doi: 10.3389/fpsyt.2014.00035. eCollection 2014. PMID 24765080
- [Background] Whitmore EA, Mikulich SK, Thompson LL, Riggs PD, Aarons GA, Crowley TJ. Influences on adolescent substance dependence: conduct disorder, depression, attention deficit hyperactivity disorder, and gender. Drug Alcohol Depend. 1997 Aug 25;47(2):87-97. doi: 10.1016/s0376-8716(97)00074-4. PMID 9298330
- [Background] Windle M. A longitudinal study of antisocial behaviors in early adolescence as predictors of late adolescent substance use: gender and ethnic group differences. J Abnorm Psychol. 1990 Feb;99(1):86-91. doi: 10.1037//0021-843x.99.1.86. PMID 2307771
- [Background] Matos M, Torres R, Santiago R, Jurado M, Rodriguez I. Adaptation of parent-child interaction therapy for Puerto Rican families: a preliminary study. Fam Process. 2006 Jun;45(2):205-22. doi: 10.1111/j.1545-5300.2006.00091.x. PMID 16768019
- [Background] Park CL, Groessl E, Maiya M, Sarkin A, Eisen SV, Riley K, Elwy AR. Comparison groups in yoga research: a systematic review and critical evaluation of the literature. Complement Ther Med. 2014 Oct;22(5):920-9. doi: 10.1016/j.ctim.2014.08.008. Epub 2014 Sep 4. PMID 25440384
- [Background] Luu K, Hall PA. Hatha Yoga and Executive Function: A Systematic Review. J Altern Complement Med. 2016 Feb;22(2):125-33. doi: 10.1089/acm.2014.0091. Epub 2015 Sep 23. PMID 26398441
- [Background] Clerkin SM, Marks DJ, Policaro KL, Halperin JM. Psychometric properties of the Alabama parenting questionnaire-preschool revision. J Clin Child Adolesc Psychol. 2007 Mar;36(1):19-28. doi: 10.1080/15374410709336565. PMID 17206878
- [Background] Barroso NE, Hungerford GM, Garcia D, Graziano PA, Bagner DM. Psychometric properties of the Parenting Stress Index-Short Form (PSI-SF) in a high-risk sample of mothers and their infants. Psychol Assess. 2016 Oct;28(10):1331-1335. doi: 10.1037/pas0000257. Epub 2015 Nov 23. PMID 26595220
- [Background] Cunningham CE, Boyle MH. Preschoolers at risk for attention-deficit hyperactivity disorder and oppositional defiant disorder: family, parenting, and behavioral correlates. J Abnorm Child Psychol. 2002 Dec;30(6):555-69. doi: 10.1023/a:1020855429085. PMID 12481971
- [Background] Kempes M, Matthys W, de Vries H, van Engeland H. Reactive and proactive aggression in children--a review of theory, findings and the relevance for child and adolescent psychiatry. Eur Child Adolesc Psychiatry. 2005 Feb;14(1):11-9. doi: 10.1007/s00787-005-0432-4. PMID 15756511
- [Background] Martinez KG, Franco-Chaves JA, Milad MR, Quirk GJ. Ethnic differences in physiological responses to fear conditioned stimuli. PLoS One. 2014 Dec 12;9(12):e114977. doi: 10.1371/journal.pone.0114977. eCollection 2014. PMID 25501365
- [Background] Milad MR, Wright CI, Orr SP, Pitman RK, Quirk GJ, Rauch SL. Recall of fear extinction in humans activates the ventromedial prefrontal cortex and hippocampus in concert. Biol Psychiatry. 2007 Sep 1;62(5):446-54. doi: 10.1016/j.biopsych.2006.10.011. Epub 2007 Jan 9. PMID 17217927
- See also: The American Academy of Child and Adolescent Psychiatry, all rights reseved. (2009). ODD A Guide for Families by the American Academy of Child and Adolescent Psychiatry. Retrieved 2018, from — https://www.aacap.org/App_Themes/AACAP/docs/resource_centers/odd/odd_resource_center_odd_guide.pdf
- See also: Lange, K.M., Maluska-Gertruda, E., Hauser, J., Reissma, A., Kauzinger, I., Tucha, L., … & Lange, K.W. (2014). Yoga and the therapy of children with attention deficit hyperactivity disorder. Yoga & Physical Therapy, 4(3), 1000168. — https://epub.uni-regensburg.de/31378/1/yoga-and-the-therapy-of-children-with-attention-deficit-hyperactivity-disorder-2157-7595.1000168.pdf
- See also: Hinshaw, S.P., & Lee, S.S. (2003). Conduct and oppositional defiant disorders. In E.J. Mash & R.A. Barkley (Eds.), Child psychopathology (3rd ed, pp. 144-198). New York: Guilford Press. — https://citeseerx.ist.psu.edu/document?repid=rep1&type=pdf&doi=8485d42325546c5fc46e2bb1e94130233fb81dc4#page=157
- See also: Psychometric properties of the Alabama parenting questionnaire-preschool revision (APQ-Pr) in 3 year-old Spanish preschoolers. Journal of Child and Family Studies, 23(5) — https://search.ebscohost.com/login.aspx?direct=true&profile=ehost&scope=site&authtype=crawler&jrnl=10621024&AN=96324836&h=mdQfC4%2FIzXPCjuK6ZdLpTglP4PqgCkMPUXbdxmMcYoPaBoXq8EK6L2nPQIJFmT3Z6LDoFUKX%2BglxuuBg14Cmig%3D%3D&crl=f
- See also: Domenech Rodríguez, M. M., Franceschi Rivera, N., Sella Nieves, Z., & Félix Fermín, J. (2013). Parenting in Puerto Rican families: Mothers and father's self-reported practices. Interamerican Journal of Psychology, 47(2). — https://www.redalyc.org/pdf/284/28430082014.pdf
- See also: Abidin, R. R. (1990). Parenting stress index-short form (p. 118). Charlottesville, VA: Pediatric Psychology Press. — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Abidin%2C+R.+R.+%281990%29.+Parenting+stress+index-short+form+%28p.+118%29.+Charlottesville%2C+VA%3A+Pediatric+Psychology+Press.&btnG=
- See also: Johnston, C., & Mash, E. J. (1989). A measure of parenting satisfaction and efficacy. Journal of clinical child psychology, 18(2), 167-175 — https://psych-parentinglab.sites.olt.ubc.ca/files/2018/02/PSOC-Johnston-and-Mash.pdf
- See also: QuickFacts. (n.d.). Retrieved January, 2018, from — https://www.census.gov/quickfacts/PR